CLINICAL TRIAL: NCT07268443
Title: Evaluation of Temporomandibular Joint With Cone-Beam Computarized Tomography at Pediatric Patients With Anterior Tooth Fracture After Trauma: A Retrospective Study
Brief Title: The Influence of Pediatric Dental Trauma on Temporomandibular Joint Disorders: A Retrospective Clinical and Radiological Analysis
Acronym: DentTraumaTMJ
Status: Completed | Type: Observational
Sponsor: Dicle University (Other)
Responsible Party: Principal Investigator, İsmet Rezani Toptancı, Asisst. Prof., Dicle University
Other Study IDs: Ethical Comitee:03.05.2012-567
Record Dates: First submitted 2025-09-09; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Evaluation of TMJ With CBCT in Pediatric Trauma Patients; Temporomandibular Joint Disorders; Dental Trauma; Anterior Teeth Fracture
Keywords: Temporomandibular disorders; CBCT analysis; Pediatric TMJ Dysfunction; Dental Trauma
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Trauma-associated TMD: Cohort: Pediatric patients aged 11-16 who presented within 1 month after complicated crown-root fractures and reported TMJ pain. CBCT and standardized clinical pain assessments were reviewed retrospectively. (n=42)
- Orthodontic Controls: Cohort Description: "Orthodontic patients aged 12-16 (Class I malocclusion) without TMJ-related complaints; pre-treatment CBCTs reviewed retrospectively under the same imaging/assessment protocol. (n=25)"

SUMMARY:
This retrospective study received ethical approval from the Ethics Committee of Dicle University Faculty of Medicine, Diyarbakır, Turkey (Decision No:03.05.2012-567). A priori power analysis (Cohen's d = 0.5, α = 0.05, 80% power) indicated that a minimum of 33 participants was required to achieve statistical reliability. Group 1 (Study Group) included 42 pediatric patients (17 females, 25 males; mean age: 12.54 ± 1.74 years) who experienced complicated crown-root fractures due to dental trauma between 2008 and 2023. All presented within one month of trauma, ensuring diagnostic uniformity. Group 2 (Control Group) included 25 orthodontic patients (9 females, 16 males; mean age: 12.60 ± 1.04 years) with Class I malocclusion and no TMJ (Temporomandibular Joint)-related symptoms. Controls were selected from orthodontic records based on skeletal harmony and availability of pre-treatment CBCT (Cone Beam Computerized Tomography) scans. In the study group, CBCT was utilized for diagnostic purposes to evaluate post-traumatic TMJ changes, as conventional imaging may not reveal subtle or asymptomatic alterations, particularly in growing children. CBCT scans in the control group were retrospectively analyzed from orthodontic records. These scans had been acquired prior to orthodontic treatment planning in accordance with standard clinical indications. In both groups, no additional radiation exposure was introduced for research purposes. Imaging followed the ALADA ( As Low As Diagnostically Acceptable) principle to balance diagnostic efficacy and radiation safety. Parental informed consent was obtained at the time of initial treatment. Data were extracted from standardized clinical and radiological records. All patients in Group 1 were evaluated and treated by a single clinician; likewise, control group patients were examined by a single orthodontist to maintain procedural consistency. All subjects underwent comprehensive clinical and CBCT-based assessments. TMJ pain was evaluated through palpation and mandibular movement (opening and closing). A four-point ordinal scale was used: No Pain, Mild, Moderate, Severe. Pain location was classified as: No Pain, Right TMJ, Left TMJ, or Bilateral. This classification supported both qualitative and quantitative assessment of TMJ symptom distribution. All CBCT scans were performed using an ICAT 3D system (Model 17-19, Imaging Sciences International, Hatfield, PA) with a 360° rotation, 120 kV, 5.0 mA, 9.6 s scan duration, and a voxel resolution of 0.3 mm. Images were analyzed using I-CAT software. The Ikeda and Kawamura (2009) method was used to measure anterior, superior, and posterior joint spaces between the condyle and glenoid fossa. The True Horizontal Line (THL) served as a reproducible reference plane. Measurements were performed with the mandible in a closed rest position. Non-parametric Mann-Whitney U tests were used for intergroup comparisons of joint space dimensions. Chi-square tests were used for categorical pain scores. A significance threshold of p ≤ 0.05 was set. Statistical analyses were performed using SPSS v21.0 (IBM Corp., Armonk, NY, USA).

DETAILED DESCRIPTION:
Introduction:

Temporomandibular disorders (TMDs) encompass a range of pathological conditions affecting the temporomandibular joint (TMJ) and related structures, with a notably high incidence in children and adolescents that increases with age. While the overall prevalence in pediatric populations is estimated at around 16%, it is significantly lower among children under ten years old. Trauma-particularly from falls or direct impacts to the jaw-is a major initiating factor, often causing acute TMD that may progress to chronic dysfunction. In children, post-traumatic pain assessment is challenging due to difficulties in localizing or describing discomfort, making early diagnosis more complex. The orofacial region's dense sensory and motor innervation adds to the complexity of TMD-related pain. These disorders primarily affect the masticatory muscles and/or TMJ, with their onset and progression influenced by initiating, predisposing, and sustaining factors. Mandibular trauma frequently involves the condylar region, further complicating functional outcomes. Currently, no single gold standard exists for comprehensive TMJ assessment, particularly in cases of direct trauma. Clinical evaluation should emphasize non-invasive, standardized protocols such as joint auscultation, palpation for pain, assessment of maximum painless mouth opening, and evaluation of mandibular lateral and protrusive movements. Pain scoring during these assessments can provide valuable insights into functional abilities. Radiological imaging is essential for diagnosis, with modalities including panoramic radiography, CT, MRI, ultrasound, and cone-beam computed tomography (CBCT). CBCT offers high-resolution, three-dimensional imaging with lower radiation doses compared to conventional CT, enabling precise measurement of condylar morphology, joint space, and structural changes. It is especially effective in detecting erosive alterations and evaluating TMJ biomechanics. Standardized CBCT protocols enhance diagnostic consistency across clinical settings. Clinically, TMDs are characterized by orofacial pain, restricted or asymmetrical jaw movement, and joint sounds during function-symptoms that can impair speech, mastication, swallowing, and overall quality of life. Physical examination may be complemented by tools such as pressure algometry, which objectively quantifies muscle tenderness; however, it is most effective when used in conjunction with other diagnostic methods. This retrospective study investigates structural and symptomatic TMJ alterations in pediatric patients with a history of dental trauma by integrating clinical findings with CBCT-based joint space measurements. An orthodontically balanced control group was included for comparison. By correlating morphometric CBCT data with clinical symptoms-an approach rarely applied systematically in pediatric trauma-the study underscores the importance of early detection, timely intervention, and preventive strategies to mitigate long-term functional impairment in growing patients.

Material and Methods:

This retrospective study was approved by the Ethics Committee of Dicle University Faculty of Medicine, Diyarbakır, Turkey (Decision No: Ethical Comitee: 03.05.2013/576). A priori power analysis was conducted using G*Power software, assuming a medium effect size (Cohen's d = 0.5), 80% statistical power, and a significance level of 0.05 (α = 0.05), indicating a minimum sample size of 33 participants to achieve statistical validity. The study group (Group 1) included 42 pediatric patients (17 females, 25 males; mean age: 12.54 ± 1.74 years) who were diagnosed with complicated crown-root fractures resulting from dental trauma between 2008 and 2023. Inclusion was restricted to cases presenting within one month post-trauma to ensure diagnostic consistency and minimize bias related to healing. All patients exhibited similar trauma severity, thereby maintaining sample homogeneity. Clinical records were reviewed to extract data on trauma-related symptoms and the presence of spontaneous jaw pain. In this cohort, cone-beam computed tomography (CBCT) was employed as a diagnostic necessity to evaluate potential temporomandibular joint (TMJ) alterations secondary to trauma. Given the limitations of clinical examination in detecting subclinical or asymptomatic TMJ changes-especially in children undergoing craniofacial development-CBCT offered a three-dimensional assessment of joint morphology to support accurate diagnosis and treatment planning. As noted by Tomina et al. CBCT offers superior 3D visualization of the condylar-glenoid fossa and is valuable for pediatric TMJ evaluation under proper clinical indications. In this study, CBCT allowed detection of displacements or trauma-related asymmetries not visible with conventional imaging. Group 2 (Control Group) consisted of 25 pediatric patients (9 girls and 16 boys) with a mean age of 12.60 ± 1.04 years. These patients exhibited no symptoms of temporomandibular joint pain. They were selected retrospectively from the records of individuals who presented to the Orthodontic Clinic for Class I orthodontic treatment between 2008 and 2023. The control group consisted of Class I malocclusion patients without TMJ symptoms, selected based on their skeletal harmony and the availability of diagnostic CBCT data. This group was chosen as a suitable clinical baseline for structural comparison instead of being a random sample of the general population. CBCT scans in the control group were not acquired for this study but retrospectively analyzed from orthodontic records. In Class I malocclusion cases, CBCT is often clinically indicated when conventional imaging is inadequate for evaluating craniofacial symmetry or TMJ morphology. Thus, no additional radiation was administered for research purposes. Following the ALADA (As Low As Diagnostically Acceptable) principle, CBCT imaging was used only when clinically justified, ensuring optimal image quality for accurate assessment while reducing radiation exposure in both the study and control groups. Informed consent was obtained from the patients' parents at the time of their initial treatment. The data used in this study were derived from patient examination forms completed during the initial assessment and follow-up forms recorded after treatment. In the study group, patient data had been previously collected by a single clinician to ensure standardization in data collection and treatment procedures. Similarly, the control group consisted of patients treated by a single orthodontist, maintaining consistency in patient selection and evaluation. In addition, all participants underwent comprehensive physical, oral, and radiological examinations as documented in their clinic records. Pain assessment occurred during palpation and mandibular movements (opening and closing). Palpation involved applying pressure to the temporomandibular joint (TMJ) area with both hands while facing the patient. Pain scoring was determined by the side of the joint where the patient felt discomfort. Pain levels were recorded using a standard pain scale to assess changes before and after treatment. For palpation and mandibular movements, pain intensity was scored using a four-level classification system: No Pain, Mild Pain, Moderate Pain, and Severe Pain. The area of joint pain was classified into four categories: No Pain, Pain in the Right TMJ, Pain in the Left TMJ, and Bilateral Pain. This scoring system allowed for the assessment of TMJ involvement and facilitated comparisons of pain distribution among participants. Cone-beam computed tomography (CBCT) was used for radiological evaluation to assess structural changes in the TMJ, providing detailed imaging of joint morphology and potential trauma-related alterations. CBCT images were obtained and evaluated before and after dental trauma treatment. In Group 2, CBCT images were obtained before treatment for patients with Class 1 orthodontic anomalies to ensure that previous interventions did not influence the assessment. In patients from group 2, evaluation was made only on CBCT images taken before the initiation of orthodontic treatment. All images in Group 1 and Group 2 were acquired using an ICAT 3D imaging system (I-CAT, Model: 17-19, Imaging Sciences International, Hatfield, PA). The scans were obtained through a 360-degree rotation at 120 kV, 5.0 mA, and a scanning duration of 9.6 seconds, with a voxel size of 0.3 mm. Image analysis was conducted using the proprietary software from I-CAT. Following the methodology described by Ikeda and Kawamura (2009), predefined anatomical landmarks were identified, and linear measurements were conducted to assess the condylar-glenoid fossa gap. The True Horizontal Line (THL) served as the reference plane for measurement. The criteria for measurement included evaluating the distances between the medial wall of the glenoid fossa and the outer side of the condyle at three specific points (anterior, superior, and posterior), while the mandible was in a closed rest position. The superior joint space was defined as the distance from the superior condylar point to the superior aspect of the glenoid fossa along the THL. Likewise, the anterior and posterior joint spaces were established by measuring the distances from the anterior and posterior condylar points to their respective aspects of the glenoid fossa. Statistical analyses were conducted to evaluate differences in joint space measurements and pain scores both within and between groups. The Mann-Whitney U test was utilized for comparisons of joint space measurements both within and among groups. For categorical pain score comparisons, the Chi-Square test was used. In this study, a p-value of ≤0.05 was considered statistically significant. All statistical analyses were performed using the SPSS software package (Version 21.0, IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria:

* Children/adolescents aged 11-16 years.
* Cases: History of complicated crown-root fracture due to dental trauma; presentation within 1 month after trauma; documented TMJ pain (palpation and/or movement); CBCT available for TMJ assessment.
* Controls: Orthodontic patients (Class I) aged 12-16 years with no TMJ-related complaints; pre-treatment CBCT available.
* Availability of standardized clinical records (pain side/intensity; mandibular movement) sufficient for retrospective analysis.
* Parental/guardian consent obtained at initial treatment per institutional policy.

Exclusion Criteria:

* Systemic/rheumatologic or neuromuscular disorders affecting the TMJ (e.g., JIA).
* Craniofacial syndromes, prior TMJ surgery, mandibular fractures involving the condyle, or forced/intubation trauma unrelated to dental injury.
* Prior or ongoing occlusal splint/orthodontic therapy likely to alter TMJ loading before baseline imaging.
* Inadequate/incomplete clinical records or poor-quality CBCT precluding reliable joint-space measurement.
* Repeated or multiple traumas where timing cannot be ascertained relative to imaging.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Single-center pediatric cohort drawn from dental trauma cases (presenting ≤1 month post-injury) and orthodontic records (Class I, asymptomatic) at a university clinic; retrospective review period 2008-2023.
  TMJ joint-space metrics via CBCT (Ikeda & Kawamura method); pain scored on a 4-point ordinal scale; ALADA principles applied; no additional radiation for research.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-06-03 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in TMJ Joint Space Measurements | Baseline CBCT (pre-treatment, obtained within 1 month after trauma) and post-treatment CBCT (performed after completion of dental/orthodontic management, up to 1 month follow-up)
  Cone-beam computed tomography (CBCT) images were obtained with patients positioned in a standardized closed-mouth rest position. Linear joint space measurements were taken between the mandibular condyle and the glenoid fossa at three reference points: anterior, superior, and posterior. The analysis followed the standardized method of Ikeda & Kawamura (2009), in which the True Horizontal Line (THL) is used as a reproducible reference plane. Measurements were recorded in millimeters directly on axial and sagittal CBCT slices using validated I-CAT software tools, ensuring high reproducibility and diagnostic accuracy. This approach minimizes positional variability and provides a reliable assessment of TMJ morphology in pediatric patients

SECONDARY OUTCOMES:
Change in TMJ Pain Intensity | Baseline (pre-treatment, within 1 month after trauma) and post-treatment (after clinical management, up to 1 month follow-up)
  Temporomandibular joint (TMJ) pain intensity was assessed using a standardized four-point ordinal scale (No pain, Mild, Moderate, Severe). Clinical evaluation included both digital palpation of the TMJ region and assessment during mandibular opening and closing movements. Pain scores were extracted from standardized clinical records and provide a reproducible measure of symptom severity in pediatric patients following dental trauma. This outcome reflects both static and functional aspects of TMJ-related discomfort.
Change in TMJ Pain Location | Baseline (pre-treatment, within 1 month after trauma) and post-treatment (after clinical management, up to 1 month follow-up)
  Pain location was evaluated by standardized clinical examination and categorized as no pain, right TMJ, left TMJ, or bilateral involvement. Classification was based on clinical records obtained during routine diagnostic visits. This approach allows qualitative assessment of the distribution of TMJ-related symptoms in pediatric patients following trauma
Change in TMJ Pain on Palpation | Baseline (pre-treatment, within 1 month after trauma) and post-treatment (after clinical management, up to 1 month follow-up)
  MJ pain was assessed by bilateral finger palpation of the joint area during clinical examination. Pain intensity was graded using a four-point ordinal scale (No pain, Mild, Moderate, Severe) and documented in standardized records. This method provides reproducible assessment of joint tenderness in children and adolescents
Change in TMJ Pain During Mandibular Movements | Baseline (pre-treatment, within 1 month after trauma) and post-treatment (after clinical management, up to 1 month follow-up)
  Functional TMJ pain was assessed during mandibular opening and closing movements. Pain intensity was scored on a four-point ordinal scale (No pain, Mild, Moderate, Severe). This outcome captures the dynamic, functional impact of trauma on TMJ activity.

OTHER OUTCOMES:
Reduction in Overall Functional Pain | Baseline (pre-treatment, within 1 month after trauma) and post-treatment (after clinical management, up to 1 month follow-up)
  Functional TMJ pain was assessed during mandibular opening and closing movements. Pain intensity was scored on a four-point ordinal scale (No pain, Mild, Moderate, Severe). This outcome captures the dynamic, functional impact of trauma on TMJ activity.

CONTACTS AND LOCATIONS:
Overall Officials: Ismet R TOPTANCI, PhD/ Assist.Prof. Dr., Study Director — Dicle Universty Dentistry Faculty Department of Pediatric Dentistry
Locations (1):
- Dicle University Faculty of Dentistry, Diyarbakır, Turkey, Diyarbakır, Sur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This is a retrospective observational study. Individual participant data will not be shared.

REFERENCES:
- [Result] Ikeda K, Kawamura A. Assessment of optimal condylar position with limited cone-beam computed tomography. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):495-501. doi: 10.1016/j.ajodo.2007.05.021. PMID 19361736
- [Result] Spinas E, Giannetti L, Mameli A, Re D. Dental injuries in young athletes, a five-year follow-up study. Eur J Paediatr Dent. 2018 Sep;19(3):187-193. doi: 10.23804/ejpd.2018.19.03.4. PMID 30063149
- [Result] Al-Khotani A, Naimi-Akbar A, Albadawi E, Ernberg M, Hedenberg-Magnusson B, Christidis N. Prevalence of diagnosed temporomandibular disorders among Saudi Arabian children and adolescents. J Headache Pain. 2016;17:41. doi: 10.1186/s10194-016-0642-9. Epub 2016 Apr 22. PMID 27102118